CLINICAL TRIAL: NCT06948591
Title: Real World Evaluation of the Safety and Effectiveness of BioBrace® Augmentation in Anterior Cruciate Ligament (ACL) Reconstruction Procedures
Brief Title: BioBrace® Augmentation in Anterior Cruciate Ligament Reconstruction Procedures
Status: Recruiting | Type: Observational
Sponsor: CONMED Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: CSP-BB0004
Record Dates: First submitted 2025-04-18; First posted 2025-04-29 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-04

CONDITIONS: ACL Tears
Keywords: ACL reconstruction; BioBrace; augmentation
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries | interventions — Anterior Cruciate Ligament Reconstruction

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- BioBrace Augment Group: An anterior cruciate ligament reconstruction is performed and BioBrace is used to augment the tissue graft.
  Interventions: Device: Anterior cruciate ligament reconstruction with BioBrace® augmentation; Procedure: Arthroscopic anterior cruciate ligament reconstruction

INTERVENTIONS:
Device: Anterior cruciate ligament reconstruction with BioBrace® augmentation — An arthroscopic anterior cruciate ligament reconstruction (ACLR) will be performed and the tissue graft will be augmented with the BioBrace® Reinforced Implant. BioBrace® is intended for use in surgical procedures for reinforcement of soft tissue where weakness exists. It is a bioresorbable, biocomposite scaffold composed of a highly porous collagen sponge and reinforced with poly-L-lactic-acid (PLLA). When used in ACLRs, it is sutured alongside the tissue graft to augment and reinforce the graft construct. BioBrace® is designed to mechanically and biologically augment weakened or torn soft tissue and can be integrated into surgeons' standard of care ACL reconstruction techniques.
Procedure: Arthroscopic anterior cruciate ligament reconstruction — An arthroscopic anterior cruciate ligament reconstruction is performed using standard surgical procedure.

SUMMARY:
This research study will evaluate mid-term clinical safety and performance outcomes of the BioBrace® Reinforced Implant when used to augment a tissue graft during anterior cruciate ligament (ACL) reconstruction.

DETAILED DESCRIPTION:
This is a multi-center, single arm, open label registry investigating anterior cruciate ligament reconstruction (ACLR) procedures where the tissue graft is augmented with BioBrace®. Subjects meeting the inclusion/exclusion criteria will be enrolled retrospectively or prospectively. Clinical evaluations will be conducted at baseline (pre-operatively) and at 6 months, 1-, 2-, and 3-years post-operatively using various patient-reported outcome measures to assess pain, function, return to activity, and safety post-surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Underwent ACL reconstruction with a tissue graft augmented with BioBrace® within the past 24 months from study start date or scheduled to undergo ACL reconstruction with a tissue graft augmented with BioBrace®.
2. Between 14 and 70 years old at the time of surgery.
3. Can understand the content of the subject information / Informed Consent Form (ICF) for the prospective portion of the study.
4. Is willing and able to participate in the prospective data collection protocol and comply with the required data collection.
5. If the subject has already undergone ACLR within the past 24 months, subject must have at least two (2) of the following measures at baseline and 1 year post-operatively:

   1. International Knee Documentation Committee (IKDC)
   2. Knee Injury and Osteoarthritis Outcome Score Junior (KOOS, JR.)
   3. Patient-Reported Outcomes Measurement Information System (PROMIS-10)
   4. Tegner Activity Scale (TAS)
   5. Anterior Cruciate Ligament - Return to Sport After Injury (ACL-RSI)
6. Positive diagnostic imaging by MRI at baseline indicating an ACL tear

Exclusion Criteria:

1. Has other concurrent medical or other conditions (chronic or acute in nature) that in the opinion of the participating investigator may prevent participation or otherwise render subject ineligible for the study.
2. Is currently participating in an investigational therapy (device and/or pharmaceutical) within 30 days prior to entering the study or such treatment is planned during the 3 years following enrollment into the study.
3. Underwent or scheduled to undergo a multi-ligament reconstruction procedure (excluding cases where a torn MCL is treated non-operatively).
4. Females of child-bearing potential who are either pregnant or breastfeeding at the time of surgery.

Ages: 14 Years to 70 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Community surrounding participating hospitals / clinics.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2025-04-08 (Actual); Primary Completion 2030-06 (Estimated); Study Completion 2030-06 (Estimated)

PRIMARY OUTCOMES:
Improvement in Function | 3 years post-op
  Improvement in function measured with International Knee Documentation Committee (IKDC) from baseline to 3 years post-surgery.
Adverse Events | Baseline, 6-months, 1-, 2-, and 3-years post-op
  Evaluation of device-related adverse events

SECONDARY OUTCOMES:
International Knee Documentation Committee (IKDC) | Baseline, 6 months, 1-, 2-years post-op
  Patient-reported functional and activity status as assessed by International Knee Documentation Committee (IKDC)
Knee Injury and Osteoarthritis Outcome Score Junior (KOOS, JR.) | Baseline, 6 months, 1-, 2-, and 3-years post-op
  Patient-reported functional and activity status as assessed by the following: Knee Injury and Osteoarthritis Outcome Score Junior (KOOS, JR.)
Patient-Reported Outcomes Measurement Information System (PROMIS-10) | Baseline, 6 months, 1-, 2-, and 3-years post-op
  Patient-reported functional and activity status as assessed by the following: Patient-Reported Outcomes Measurement Information System (PROMIS-10)
Tegner Activity Scale (TAS) | Baseline, 6 months, 1-, 2-, and 3-years post-op
  Patient-reported functional and activity status as assessed by: Tegner Activity Scale (TAS).
Anterior Cruciate Ligament - Return to Sport After Injury (ACL-RSI) | 6 months, 1-, 2-, and 3-years post-op
  Patient-reported functional and activity status as assessed by the following: Anterior Cruciate Ligament - Return to Sport After Injury (ACL-RSI)
Secondary Surgical Intervention(s) | 6 months, 1-, 2-, and 3-years post-op
  The percentage of subjects who required additional surgical procedures following discharge from the BioBrace ACLR index procedure will be reported.
Re-tear Rate | 6 months, 1-, 2-, and 3-years post-op
  Re-tear rate of the surgically reconstructed ACL tissue graft augmented with BioBrace. The percentage of subjects who experienced a re-tear of the augmented ACL tissue graft will be reported.

CONTACTS AND LOCATIONS:
Locations (1):
- ConMed, New Haven, Connecticut, United States